CLINICAL TRIAL: NCT07231510
Title: KARU-FERTIL: Chlordecone Exposure and Female Fertility
Brief Title: Chlordecone Exposure and Female Fertility
Acronym: KARU-FERTIL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Institut Pasteur de Guadeloupe (Unknown); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2023/08; 2023-A01755-40 (Registry Identifier: ANSM)
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Infertility Female
Keywords: polycystic ovarian syndrome; endometriosis; female infertility,; ovarian reserve; environmental exposures; chlordecone; kepone
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chlordecone is an organochlorine pesticide used in the French West Indies (FWI) from 1972 to 1993 to control the banana root borer. Due to its very long persistence the population continues to be exposed to this chemical through their food consumptions. Although, chlordecone have been associated in animal study impairment of ovarian reserve, to date, no study has been published concerning the link between chlordecone exposure and female fertility. The main objective of this project is to study the association between chlordecone exposure and anti-mullerian hormone (AMH) in women consulting for couple infertility in Guadeloupe.

DETAILED DESCRIPTION:
Chlordecone is an organochlorine pesticide used in the French West Indies (FWI) from 1972 to 1993 to control the banana root borer. Due to its very long persistence the population continues to be exposed to this chemical through their food consumptions. Chlordecone is an endocrine-disrupting chemical with well-defined estrogenic and progestagenic properties in vivo and in vitro. To date, no study has been published concerning the link between chlordecone exposure and female fertility. Nevertheless, mammalian studies in females have consistently reported that chlordecone exposure impairs ovulation and leads to a reduced ovarian reserve. In addition, there are questions about the impact of other environmental exposures, including by non-targeted approaches, and also of the vaginal and endometrial microbiome on female fertility.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18 to 39 years
* Consulting for couple infertility at the Centre Caribéen de Médecine de la Reproduction (CCMR, Caribbean Center for Reproductive Medicine) of the University Hospital of Guadeloupe
* Free, informed and written consent

Exclusion Criteria:

* Women aged from 18 to 39 years
* Consulting for couple infertility at the Centre Caribéen de Médecine de la Reproduction (CCMR, Caribbean Center for Reproductive Medicine) of the University Hospital of Guadeloupe
* Free, informed and written consent

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women consulting for couple infertility in Guadeloupe.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2028-01-26 (Estimated)

PRIMARY OUTCOMES:
Levels of AMH according to terciles of chlordecone levels. | AMH levels will be measured during the assessment conducted for assisted reproductive technology (ART) and will date from less than one year before inclusion
  The purpose is to study the association between chlordecone exposure and AMH levels in women consulting for couple infertility in Guadeloupe.

SECONDARY OUTCOMES:
Number of antral follicles according to terciles of chlordecone levels. | between days 2 and 4 of the spontaneous menstrual cycle
  Transvaginal ultrasound for antral follicle count will be performed between days 2 and 4 of the spontaneous menstrual cycle, the number of antral follicles corresponds to the total number of antral follicles in both ovaries, with a diameter between 2 and 10 mm.
AMH levels and antral follicle count according to the levels of other POPs | baseline
  AMH levels and antral follicle count
relationship between exposure to chlordecone and other POPs and the risk of the main causes of female infertility | baseline
  main causes of female infertility : Endometriosis ; Polycystic ovary syndrome (PCOS) ; Decreased ovarian reserve
Chlordecone levels according to the outcomes of IVF/ICSI management: | changes from baseline to 2 years after
  relationship between occupational exposure to solvents and others factors described :
  * Endometrial thickness,
  * Peak estraiol,
  * Number of oocytes collected,
  * Number of mature oocytes collected,
  * Number of zygotes,
  * Embryo quality,
  * Blastocyst number,
  * Number of frozen embryos,
  * Biological pregnancy,
  * Clinical pregnancy,
  * Live birth.

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Garlantezec, MD PhD, Study Director — CHU de Rennes - Université de Rennes
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe